CLINICAL TRIAL: NCT06721260
Title: METRICS Study: Metabolic Evaluation Through Resting Indirect Calorimetry in Bladder Cancer
Brief Title: Metabolism Evaluation Through Resting Indirect Calorimetry in Bladder Cancer (METRICS)
Acronym: METRICS
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Jill Hamilton-Reeves, PhD RD LD, Professor, University of Kansas Medical Center
Other Study IDs: STUDY00160673
Record Dates: First submitted 2024-11-26; First posted 2024-12-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; resting energy expenditure; cachexia; growth differentiation factor 15 (GDF-15); Nutrition status; radical cystectomy; neoadjuvant chemotherapy; body composition
MeSH Terms: conditions — Urinary Bladder Neoplasms; Cachexia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is being done to learn more about energy needs and muscle function during treatment for bladder cancer. These insights can help improve future patient care. The study team found in a previous study that resting energy can be different than what estimates show. Patients with bladder cancer are known to suffer a decline in physical resilience over time. Monitoring patients to understand these changes better could help design future treatments with these vulnerabilities in mind.

DETAILED DESCRIPTION:
The investigators' long-term goal is to improve cachexia treatment for patients with cancer. The project is significant because identifying cachexia earlier in its onset allows for earlier and more successful treatment. Major barriers to early detection and treatment are: 1) clear specific lab tests to confirm the diagnosis and 2) identifying when resting energy expenditure (REE) increases. It is the investigators' expectation that at the completion of these descriptive studies, key factors will be identified to guide earlier detection and treatment of cachexia. Platinum-based chemotherapy and surgery are a dual-phase treatment regimen to treat bladder cancer that has a high risk of worsening cachexia compared to other cancer types not requiring such an intensive treatment regimen. Inhibition of Growth differentiation factor 15 (GDF-15) is a promising preventive strategy against cachexia in patients with bladder cancer. Understanding GDF-15 and REE changes over the course of treatment could inform proactive rather than reactive strategies to support the health of these patients and translate to patients with other types of cancer. The objective of this application is to assess changes in GDF-15 and REE levels during the treatment course for advanced bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed cancer diagnosis
* Scheduled for platinum-based chemotherapy followed by radical cystectomy
* Adequate renal and cardiac function for platinum-based chemotherapy

Exclusion Criteria:

* Prior chemotherapy or radiotherapy for bladder cancer
* Severe cardiac, renal, hepatic, respiratory or metabolic diseases
* Pregnant or breastfeeding
* Uncontrolled conditions that could affect study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential patients will be scheduled for treatment (chemotherapy and radical cystectomy) for bladder cancer at the University of Kansas Health System.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To assess Resting Energy Expenditure (REE) changes across key treatment milestones. | From enrollment, prior to chemotherapy, to 3 weeks after radical cystectomy.
  Resting Energy Expenditure (REE) will be measured using indirect calorimetry before and after chemotherapy and radical cystectomy and will be associated with clinical outcomes.

SECONDARY OUTCOMES:
Blood biomarkers | From enrollment, prior to chemotherapy, to 3 weeks after radical cystectomy.
  Blood will be collected at study visits and growth differentiation factor-15 (GDF-15) concentration will be evaluated.
Inflammation marker | From enrollment, prior to chemotherapy, to 3 weeks after radical cystectomy.
  Blood will be collected at study visits and Interleukin-6 (IL-6) concentration will be evaluated.
Immune inflammation marker | From enrollment, prior to chemotherapy, to 3 weeks after radical cystectomy.
  Blood will be collected at study visits and tumor necrosis factor alpha (TNFa) concentration will be evaluated.
Body composition | From enrollment, prior to chemotherapy, to 3 weeks after radical cystectomy.
  Changes in muscle and fat mass will be assessed using dual-energy X-ray (DXA) at study visits.
Nutrition assessment | From enrollment, prior to chemotherapy, to 3 weeks after radical cystectomy.
  The Patient-Generated Subjective Global Assessment (PG-SGA) and 24-hour dietary recalls will be administered in an interview format by trained study personnel. These will take place at study visits.
Grip strength measurement | From enrollment, prior to chemotherapy, to 3 weeks after radical cystectomy.
  A hand dynamometer will be used to measure grip strength at study visits.
Quality of Life (QOL) and Fatigue assessment | From enrollment, prior to chemotherapy, to 3 weeks after radical cystectomy.
  FACIT-Fatigue questionnaires will be administered to evaluate changes in health-related quality of life (HRQOL) at study visits.
Quality of Life (QOL) during bladder cancer treatment assessment | From enrollment, prior to chemotherapy, to 3 weeks after radical cystectomy.
  FACT-Bl-Cys questionnaires will be administered to evaluate changes in health-related quality of life (HRQOL) at study visits.

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Hamilton-Reeves, PhD, RD, CSO, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States